CLINICAL TRIAL: NCT04629989
Title: The Effects of Two Systems Above Low-flow Nasal Cannula on Arterial Oxygen Tension in Patients With COVID-19 : Surgical Face Mask Versus Double-trunk Mask
Brief Title: Comparison of the Surgical Facemask With the Double-trunk Mask on Oxygenation in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Poncin, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DTM-003
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Hypoxemia
Keywords: Double-Trunk Mask; Surgical Mask
MeSH Terms: conditions — COVID-19; Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-flow nasal cannula (Active Comparator): The standard oxygen delivery system (low-flow nasal cannula) is worn by the patient, without the DTM or the SM
  Interventions: Other: Standard Oxygen Delivery System
- Double-Trunk Mask (Experimental): The Double-Trunk Mask is placed above the standard oxygen delivery system (low-flow nasal cannula).
  Interventions: Other: Double-Trunk Mask
- Surgical Mask (Experimental): The Surgical Mask is placed above the standard oxygen delivery system (low-flow nasal cannula).
  Interventions: Other: Surgical Mask

INTERVENTIONS:
Other: Standard Oxygen Delivery System — The standard oxygen delivery system (low-flow nasal cannula or oxygen mask) is worn by the patient for 1 hour.
  Arms: Low-flow nasal cannula
Other: Double-Trunk Mask — The Double-Trunk Mask above the standard oxygen delivery system (low-flow nasal cannula or oxygen mask) is worn by the patient for 1 hour.
  Arms: Double-Trunk Mask
Other: Surgical Mask — The Surgical Mask above the standard oxygen delivery system (low-flow nasal cannula or oxygen mask) is worn by the patient for 1 hour.
  Arms: Surgical Mask

SUMMARY:
This study will compare the impact of two systems above low-flow nasal cannula on the arterial oxygen tension in patients with COVID-19. The two systems are the Surgical Mask (SM) and the Double-Trunk Mask (DTM).

DETAILED DESCRIPTION:
Hospitalized patients with COVID-19 typically present with hypoxemia. In some patients, hypoxemia can be corrected with low flow nasal cannula. When placed above nasal cannula, some systems have demonstrated their interest in improving the performance of patient's oxygen delivery. For example, two recent studies have shown that adding a Double-Trunk Mask (DTM) or Surgical Mask (SM) above nasal cannula has the potential to improve the PaO2 despite no change in oxygen output (Duprez et al., J Clin Monit Comput 2020; Montiel et al., Ann Intensive Care 2020). However, there is no study comparing the relative effectiveness of these 2 systems.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive
* SpO2 between 92 and 96% with low-flow oxygen therapy
* Oxygen output at baseline between 3 and 7 L/min.

Exclusion Criteria:

* Pulmonary disease with hypercapnia
* Confusion
* Contra-indications to arterial blood gas sampling (peripheral arteriopathy, bleeding disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Changes in PaO2 | At baseline and 30 minutes after wearing the randomized oxygen delivery system
  Oxygen tension (PaO2) in mmHg will be analyzed from a sample taken from the arterial system

SECONDARY OUTCOMES:
Change in PaCO2 | At baseline and 30 minutes after wearing the randomized oxygen delivery system
  Carbon dioxide tension (PaCO2) in mmHg will be analyzed from a sample taken from the arterial system.
Change in pH | At baseline and 30 minutes after wearing the randomized oxygen delivery system
  Potential of Hydrogen (pH) will be analyzed from a sample taken from the arterial system.
Change in respiratory rate | At baseline, 30 minutes and 60 minutes after wearing the randomized oxygen delivery system
  Respiratory rate is measured during one minute by visual inspection.
Change in dyspnea | At baseline and 60 minutes after wearing the randomized oxygen delivery system
  Dyspnea is rated with a visual analogic scale (0 to 100mm).
Change in O2 output | At 30 minutes and 60 minutes after wearing the randomized oxygen delivery system
  The O2 output will be adjusted to recover the baseline SpO2 reading. The O2 output will be read from the position of the ball inside the flowmeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium